CLINICAL TRIAL: NCT03089177
Title: Community Activation for Prevention (CAPs): A Randomized Controlled Trial of Community Gardening
Brief Title: Community Activation for Prevention (CAPs): A Study of Community Gardening
Acronym: CAPs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Colorado, Boulder (Other)
Collaborators: Michigan State University (Other); Colorado School of Public Health (Other); University of South Carolina (Other); Colorado State University (Other); Denver Urban Gardens (Unknown)
Responsible Party: Principal Investigator, Jill Litt, Associate Professor, Environmental Studies, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16-0644
Record Dates: First submitted 2017-02-17; First posted 2017-03-24 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Cancer; Obesity; Lifestyle, Sedentary; Physical Activity; Health Behavior; Chronic Disease; Diet Modification
Keywords: Randomized Controlled Trial; Community Gardening; Health Behavior Change; Physical Activity; Diet; Obesity; Cancer Prevention; Neighborhood
MeSH Terms: conditions — Neoplasms; Obesity; Sedentary Behavior; Motor Activity; Health Behavior; Chronic Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Garden Intervention Group (Experimental): Participants randomized to the Community Garden Intervention Group will receive the garden intervention. Participants will be assigned a plot for one season and will receive a standard package of services and amenities to support participation in the community garden.
  Interventions: Behavioral: Community Garden Intervention
- Wait List Control Group (No Intervention): Participants randomized to the Wait List Control Group will remain on community gardening waiting lists and will not receive the garden intervention.

INTERVENTIONS:
Behavioral: Community Garden Intervention — The investigators will recruit prospective adult gardeners who have not been gardening for the past two years and who are listed on Denver Urban Gardens (DUG) wait lists. Individuals randomized to the garden intervention will receive a standardized garden resource package, which includes the following:
  1. A garden plot in a Denver Urban Garden
  2. Seeds and plant starts
  3. Introductory gardening workshop
  4. Social events including garden-specific events and garden mentoring.
  The Wait List Control group will remain on the community gardening wait lists and will not receive these resources.
  Duration of the intervention is 1 year.
  Arms: Community Garden Intervention Group

SUMMARY:
The investigators previous studies show that community gardening is associated with reduction of key health behaviors for cancer prevention in diverse populations. Community gardeners eat more fruits and vegetables per day, are more physically active, and are more likely to avoid age-associated increase in body mass index (BMI). The effect is partially explained by the finding that gardeners are more socially involved, and feel more social support than non-gardeners.

The investigators propose a randomized controlled trial to determine whether community gardening improves cancer-preventive behaviors among a multi-ethnic, low-income adult population and elucidate the pathways that shape cancer-preventive behaviors. A randomized controlled trial is needed to demonstrate that the observed behavioral differences are due to the effect of gardening as an intervention rather than self-selection by gardeners.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent in English or Spanish
* Aged 18 or over
* Currently on the wait list for a new garden
* Not have gardened in the past 2 gardening seasons

Exclusion Criteria:

* Is not able to complete the study requirements in Spanish or English
* Aged 17 or younger
* Has gardened in the past 2 gardening seasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in fruit and vegetable intake from baseline at 20 weeks and 52 weeks | Measurements will occur during weeks 1-2 (3 random recalls) and week 20 (3 random recalls) and week 48 (3 random recalls)
  9 24-hour diet recalls will be collected randomly
Change in sedentary time from baseline at 20 weeks and 48 weeks | 3 measurements over one year, T1 (week 1), T2 (week 20), T3 (week 52)
  Accelerometers will be adhered to thigh and collect data for 7 days
Change in fiber Intake from baseline at 20 weeks and 52 weeks | Measurements will occur during weeks 1-2 (3 random recalls) and week 20 (3 random recalls) and week 48 (3 random recalls)
  9 24-hour diet recalls will be collected randomly
Change in Healthy Eating Index (HEI) from baseline at 20 weeks and 52 weeks | Measurements will occur during weeks 1-2 (3 random recalls) and week 20 (3 random recalls) and week 48 (3 random recalls)
  9 24-hour diet recalls will be collected randomly
Change in moderate-to-vigorous physical activity (MVPA) from baseline to 20 weeks | 3 measurements over one year, T1 (week 1), T2 (week 20), T3 (week 52)
  Accelerometers will be adhered to thigh and collect data for 7 days
Change in waist circumference from baseline to 20 weeks and 52 weeks | 3 measurements over one year, T1 (week 1), T2 (week 20), T3 (week 52)
  Measurement of waist circumference (cm)
Change in weight (kg) from baseline to 20 weeks and 52 weeks | 3 measurements over one year, T1 (week 1), T2 (week 20), T3 (week 52)
  Objective measurement of weight will be collected

SECONDARY OUTCOMES:
Change in Perceived Stress from baseline to 20 weeks and 52 weeks | 3 measurements over one year, T1 (week 1), T2 (week 20), T3 (week 52)
  Validated scale of perceived stress will be completed

CONTACTS AND LOCATIONS:
Overall Officials: Jill S Litt, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
The investigators will store all Individual Participant Data in a HIPPA compliant database separate from the study database. All analysis will be conducted on an analytic data set, stripped of indirect and direct identifiers.

REFERENCES:
- [Derived] Coringrato E, Alaimo K, Leiferman JA, Villalobos A, Buchenau H, Decker E, Fahnestock L, Quist P, Litt JS. A process evaluation of a randomized-controlled trial of community gardening to improve health behaviors and reduce stress and anxiety. Sci Rep. 2024 Jun 13;14(1):13620. doi: 10.1038/s41598-024-63889-w. PMID 38871715
- [Derived] Alaimo K, Beavers AW, Coringrato E, Lacy K, Ma W, Hurley TG, Hebert JR. Community Gardening Increases Vegetable Intake and Seasonal Eating From Baseline to Harvest: Results from a Mixed Methods Randomized Controlled Trial. Curr Dev Nutr. 2023 Apr 15;7(5):100077. doi: 10.1016/j.cdnut.2023.100077. eCollection 2023 May. PMID 37215644
- [Derived] Litt JS, Alaimo K, Harrall KK, Hamman RF, Hebert JR, Hurley TG, Leiferman JA, Li K, Villalobos A, Coringrato E, Courtney JB, Payton M, Glueck DH. Effects of a community gardening intervention on diet, physical activity, and anthropometry outcomes in the USA (CAPS): an observer-blind, randomised controlled trial. Lancet Planet Health. 2023 Jan;7(1):e23-e32. doi: 10.1016/S2542-5196(22)00303-5. PMID 36608945
- [Derived] Villalobos A, Alaimo K, Erickson C, Harrall KK, Glueck DH, Buchenau H, Buchenau M, Coringrato E, Decker E, Fahnestock L, Hamman RF, Hebert JR, Hurley TG, Leiferman JA, Li K, Quist P, Litt JS. CAPS on the move: Crafting an approach to recruitment for a randomized controlled trial of community gardening. Contemp Clin Trials Commun. 2019 Nov 8;16:100482. doi: 10.1016/j.conctc.2019.100482. eCollection 2019 Dec. PMID 31799473
- [Derived] Litt JS, Alaimo K, Buchenau M, Villalobos A, Glueck DH, Crume T, Fahnestock L, Hamman RF, Hebert JR, Hurley TG, Leiferman J, Li K. Rationale and design for the community activation for prevention study (CAPs): A randomized controlled trial of community gardening. Contemp Clin Trials. 2018 May;68:72-78. doi: 10.1016/j.cct.2018.03.005. Epub 2018 Mar 18. PMID 29563043